CLINICAL TRIAL: NCT00542737
Title: Improving Ventilator Management and Preventing Injury to Patients With Acute Respiratory Failure
Brief Title: Evaluating a Web-Based Ventilator Management Educational Program for Clinicians (The Lung Injury Knowledge Network [LINK] Study)
Acronym: LINK
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Gordon D. Rubenfeld, MD, University of Toronto, Sunnybrook Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 518; R01HL067939 (NIH); GC1# A19846
Record Dates: First submitted 2007-10-10; First posted 2007-10-11 (Estimated); Last update posted 2013-07-11 (Estimated); Status verified 2010-08

CONDITIONS: Respiratory Distress Syndrome, Adult
Keywords: Acute Lung Injury; Acute Respiratory Distress Syndrome; Acute Respiratory Failure; Web-Based Intervention; Lung Preventive Ventilation
MeSH Terms: conditions — Respiratory Distress Syndrome; Acute Lung Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early Intervention Group (Active Comparator)
  Interventions: Behavioral: Web-Based Educational Program
- Delayed Intervention Group (Active Comparator)
  Interventions: Behavioral: Web-Based Educational Program

INTERVENTIONS:
Behavioral: Web-Based Educational Program — Participating clinicians at each hospital will access the Web site as often as necessary for a 6-month period. The Web site will contain background and educational information on ALI/ARDS and LPV, including how to recognize ALI/ARDS and how to implement LPV in patients. Scholarly articles and other materials, including a chart to help clinicians determine appropriate ventilator settings for each patient, will be available to download. Clinicians will also be able to email questions to critical care experts.

SUMMARY:
Acute lung injury/acute respiratory distress syndrome (ALI/ARDS) is a severe lung condition that causes respiratory failure. Individuals with ALI/ARDS often require the use of a respirator or artificial breathing machine, known as a mechanical ventilator, while in an intensive care unit (ICU). Research has shown that lung protective ventilation (LPV), a type of mechanical ventilation technique, is an effective way to reduce the number of deaths due to ALI/ARDS. This study will evaluate the effectiveness of a Web-based educational program that aims to educate ICU clinicians about the use of LPV in patients with ALI/ARDS.

DETAILED DESCRIPTION:
ALI/ARDS is a life-threatening condition that involves inflammation of the lungs and fluid accumulation in the air sacs, leading to low blood oxygen levels and respiratory failure. Common causes include pneumonia, septic shock, and lung trauma, and most patients require immediate care in an ICU. The main form of treatment for ALI/ARDS is the delivery of oxygen and a continuous level of pressure to the damaged lungs through mechanical ventilation. Each year, 74,500 people die due to ALI/ARDS and 22% of these deaths could be prevented with the use of LPV. LPV is a mechanical ventilation technique in which lower volumes of oxygen are administered. The purpose of this study is to implement and evaluate a Web-based educational program that will provide educational and instructional resources about ALI/ARDS and LPV to ICU clinicians, including physicians, nurses, and respiratory therapists.

Hospitals participating in this study will be randomly assigned to access the Web site at either the beginning of the study period or a later time. Participating clinicians at each hospital will access the Web site as often as necessary for a 6-month period. The Web site will contain background and educational information on ALI/ARDS and LPV, including how to recognize ALI/ARDS and how to implement LPV in patients. Scholarly articles and other materials, including a chart to help clinicians determine appropriate ventilator settings for each patient, will be available to download. Clinicians will also be able to email questions to critical care experts. At the end of the 6-month study period, study staff will compare the number of patients receiving LPV to the number of patients who received LPV prior to the start of the study.

ELIGIBILITY:
Inclusion Criteria for Hospitals:

* Between 10 and 20 ICU beds with 5 to 10 ALI/ARDS patients cared for each month
* Provide critical care services
* Keep electronic medical records on ICU patients
* ICU staff must have access to computers with Intranet or Internet

Inclusion Criteria for Clinicians:

* Provide care for mechanically ventilated patients in ICUs
* Willing to participate by viewing Web site

Exclusion Criteria for Hospitals:

* Cardiac, cardiothoracic, neurosurgical, neonatal, or pediatric ICUs
* Residents and fellows must provide care to majority of critically ill patients
* Fewer than 5 to 10 ALI/ARDS patients cared for each month

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2009-02; Primary Completion 2013-09 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Percentage of eligible patients with ALI/ARDS who are receiving LPV | Measured at Month 6

CONTACTS AND LOCATIONS:
Overall Officials: Gordon D. Rubenfeld, MD, Principal Investigator — University of Toronto, Sunnybrook Health Sciences
Locations (1):
- University of Toronto, Sunnybrook Health Sciences, Toronto, Ontario, Canada